CLINICAL TRIAL: NCT06751927
Title: Uptake of Varenicline and Strategies for Enhanced Engagement in Treatment for Smoking Cessation
Brief Title: New Strategies to Enhance Smoking Cessation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB24-1204
Record Dates: First submitted 2024-12-20; First posted 2024-12-30 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Educational Intervention (Experimental): Study participants will watch a video containing research findings related to smoking cessation and information on varenicline, a medication to help patients quit smoking.
  For participants who select varenicline and/or nicotine replacement, medications will be mailed to their residence and standard follow-up and medication support practices will be adhered to check on progress.
  Participants will be randomized to between educational intervention and usual care arm.
  Some participants who have no access to a video-enabled device or reliable internet and will provide them a tablet with broadband internet for a period of 3 months.
  Interventions: Behavioral: Educational Video
- Treatment-as-usual (TAU) (No Intervention): Treatment-as-usual (TAU) session with discussion of FDA-approved smoking medication. Treatment as usual includes discussion and facts about cessation medication options as a standard of care with a standard video on smoking cessation treatment.
  For participants who select varenicline and/or nicotine replacement, medications will be mailed to their residence and standard follow-up and medication support practices will be adhered to check on progress.
  Some participants who have no access to a video-enabled device or reliable internet and will provide them a tablet with broadband internet for a period of 3 months.
- Focus Group (No Intervention): 3 focus groups with 6-8 patients each to provide feedback on video production format and salience of relevant content

INTERVENTIONS:
Behavioral: Educational Video — Education video on smoking, nicotine receptor involvement in addiction, craving, withdrawal and mechanisms of action for nicotine replacement and varenicline.
  Arms: Educational Intervention

SUMMARY:
The study goal is to get feedback on ways researchers can communicate complex research findings on smoking cessation to better inform patients' decisions to use medication and/or quit smoking. This will help researchers and clinicians to provide effective, easy-to-implement treatments designed to address tobacco-related health disparities in Black and other racial/ethnic subgroups. It will also help improve health literacy to change misperceptions and mistrust on uptake of varenicline and other medication for quitting smoking. A professionally made video will explain research findings relevant for varenicline's mechanisms and outcomes relative to other treatment options.

There are 2 parts to this study:

* Part 1: Focus Group to help develop the educational tool intervention
* Part 2: Randomized portion of study. In this part of the study, participants will be randomized (like flip of coin) to take part in receive the experimental educational intervention or usual methods to help stop smoking. Participants in either arm can choose to receive varenicline and it will be provided as part of study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must smoke at least 10 cigarettes/day and do not currently use a smoking cessation medication.
* Ages 18-75.
* Agree to complete surveys and measures within study.
* Ability to understand English and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who are receiving any other smoking cessation medications.
* Patients who are pregnant and/or lactating.
* Patients with psychiatric contraindications that can prevent adherence to protocol or use of intervention tools in study. For inclusivity on trial, psychiatric contraindications and ability for patient to participate in trial will be assessed on an individual basis by study investigator.
* Patients who have a contraindication with varenicline.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2025-04-24 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Acceptability of the experimental video intervention | 24 weeks
  This will be assessed using a modified version of the Client Satisfaction Questionnaire which assesses items such as quality, effectiveness, and intrusiveness on the 10-point Likert scale (0=not at all, 10=very much).
Determine whether provision of technology access and support will improve program attendance and smoking outcomes | 24 weeks
  This will be assessed using a modified version of the Client Satisfaction Questionnaire specific to technology component which assesses items such as quality, effectiveness, and intrusiveness on the 10-point Likert scale (0=not at all, 10=very much).
Trial feasibility | End of study recruitment (6 months)
  ability to enroll and follow-up with the planned number of participants within the specified time frame.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea C. King, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Are the UChicago researchers conducting this study or any portion of the study at a non-UChicago site ? NO